CLINICAL TRIAL: NCT07211646
Title: The Assessment of Human Sleep and Its Functions
Acronym: SS_Sleep
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: StimScience Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 19042
Record Dates: First submitted 2025-09-23; First posted 2025-10-08 (Actual); Last update posted 2025-10-08 (Actual); Status verified 2025-09

CONDITIONS: Insomnia
Keywords: tES intervention for Sleep
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Intervention Model Description: Participants randomly get control or sham, vs. stimulation variations
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- tES Stimulation (Experimental): Within person group to test different interventions in randomized order
  Interventions: Other: sham tES; Other: Fixed tES; Other: Personalized tES

INTERVENTIONS:
Other: sham tES — short 30s sham stimulation
Other: Fixed tES — Fixed stimulation parameters for all participants
Other: Personalized tES — Stimulation parameters personalized for each participant

SUMMARY:
The purpose of this study is to look at the effects of targeted brain stimulation when falling asleep and on sleep quality.

DETAILED DESCRIPTION:
The purpose of this study is to see the effects of targeted brain stimulation when falling asleep and on sleep quality. The study uses non-invasive Transcranial Electrical Stimulation (tES), and/or a standard electroencephalogram (EEG). We may also measure eye movements, muscle activity, and heart rhythm. We may play audio during the stimulation.

The sessions can include full overnight sleep or short nap session.

ELIGIBILITY:
Inclusion Criteria:

* 18-75 year olds

Exclusion Criteria:

* Epilepsy
* Seizure History
* Serious head injury or brain surgery
* Migraines
* Metal implants in head
* Pacemaker or implanted devices
* Pregnancy
* Any serious medical condition other than insomnia

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2019-05-20 (Actual); Primary Completion 2028-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Sleep Efficiency Change | up to 6 weeks
  Sleep efficiency (time slept as a percentage time spent in bed) changes across the different interventions for each subject and aggregate that across subjects
Sleep Onset Change | 1 day to 6 weeks
  Changes in time to fall asleep across the different interventions for each subject and aggregate that across subjects

CONTACTS AND LOCATIONS:
Locations (1):
- StimScience, Berkeley, California, United States